CLINICAL TRIAL: NCT05877274
Title: Sodium Channel Mutations (SCN9A, SCN10A) in the Anterior Cutaneous Nerve Entrapment Syndrome (ACNES)
Brief Title: Sodium Channel Mutations in Patient With the Anterior Cutaneous Nerve Entrapment Syndrome (ACNES)
Acronym: Nav-ACNES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maxima Medical Center (Other)
Responsible Party: Principal Investigator, dr. RMH Roumen, surgeon, Head of surgery, Principal Investigator, Maxima Medical Center
Other Study IDs: NL84021.015.23
Record Dates: First submitted 2023-04-16; First posted 2023-05-26 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-05

CONDITIONS: Anterior Cutaneous Nerve Entrapment Syndrome; Nerve Entrapment Syndrome; Chronic Pain Syndrome
Keywords: ACNES; Sodium channel mutations
MeSH Terms: conditions — Charcot-Marie-Tooth Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — One whole blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with ACNES: Patients with ACNES who fulfill the inclusion criteria.
  Interventions: Other: Sodium channel mutation

INTERVENTIONS:
Other: Sodium channel mutation — Mutation of the genes SCN9A and SCN10A, which encode for Sodium channel 1.7 and 1.8.

SUMMARY:
The goal of this observational study is to learn about sodium channel (Nav) mutations in patients with the Anterior Cutaneous Nerve Entrapment Syndrome (ACNES). This study will give more insight into the pathophysiology of ACNES, which is still largely unknown.

The primary objective is to determine if there are mutations of Nav1.7 and Nav1.8 in patients with ACNES. Therefore, one blood sample will be drawn, in which the mutations will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must be diagnosed with ACNES and receive treatment at our outpatient clinic. Additionally, subject has to meet one of the following criteria:

* Known to have a first- or second-degree relative with ACNES;
* Have more than one recurrence of ACNES after a pain free period or ACNES at multiple locations in the abdominal wall;
* Persistent pain after posterior neurectomy.

Exclusion Criteria:

* Inability to understand Dutch language.
* Known neuromuscular or neurodegenerative disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are diagnosed with ACNES and receive treatment at our outpatient clinic, and fulfill the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Sodium Channel 1.7 and 1.8 mutation. | Blood samples for SCN analysis will be taken only once after obtaining informed consent. This is the start of the study. Outpatient discharge (free of pain or no treatment options) is end of study. Treatment period can be a couple of weeks or months.
  Number of SCN9A and SCN10A mutations. Each mutation will be classified following one of three classes; unknown pathogenicity, probable pathogenicity, and pathogen variant.

SECONDARY OUTCOMES:
Correlation between mutations and known cause of ACNES. | Baseline data will be obtained during first outpatient visit, before start of the treatment. The first outpatient visit takes 30 minutes (standard of care).
  Patients are asked (standard of care) if there is a possible cause of the ACNES. Correlations between the causes of ACNES and any identified mutations will be examined.
Correlation between mutations and pain score at start of treatment. | Baseline data will be obtained during first outpatient visit, before start of the treatment. The first outpatient visit takes 30 minutes (standard of care).
  Patients are asked (standard of care) about the average pain score following the 0-10 numeric rating scale (NRS) (0 = no pain, 10 worst possible pain).
  Correlations between the NRS pain score and found mutations will be examined.
Correlation between mutations and treatment response. | Treatment response will be assessed after each treatment during the treatment period at our outpatient clinic, up to 6 weeks after treatment.
  Patients follow different treatments according standard of care for ACNES. Starting with trigger point injections with a local anesthetic, if this treatment is not sufficient, it is followed by Pulse Radiofrequency. When patients still experience pain after minimal invasive treatments, a surgical neurectomy is performed.
  Correlations between treatment outcome after the different treatment options and found mutations will be examined. Treatment is defined successful if the patient does not need additional treatment, has >50% pain reduction, or reduction of >4 NRS points.

CONTACTS AND LOCATIONS:
Overall Officials: Rudi Roumen, MD, PhD, Principal Investigator — Maxima Medical Center
Locations (1):
- Maxima Medical Center, Veldhoven, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided